CLINICAL TRIAL: NCT05458310
Title: The Development of Incisional Hernia in Relation to Specimen Extraction Site After Laparoscopic Colorectal Surgeries: A Retrospective Single Centered Cohort Study
Brief Title: The Development of Incisional Hernia in Relation to Specimen Extraction Site After Laparoscopic Colorectal Surgeries
Status: Completed | Type: Observational
Sponsor: Prince Sultan Military College of Health Sciences (Other)
Responsible Party: Principal Investigator, Faisal Alboqami, Resident General Surgery, Prince Sultan Military College of Health Sciences
Other Study IDs: HP-01-R-079
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospec/ve cohort study of colon cancer patients who underwent laparoscopic colorectal surgeries at Prince Sultan Military Medical City (PSMMC) in Riyadh, Saudi Arabia. The aim of this study is to determine the best site for specimen extrac/on with lowest risk of developing incisional hernia a0er laparoscopic colorectal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* The study included all colorectal cancer patients over 2 years who were followed up or admitted to PSMMC under the service of colorectal surgery unit and who underwent laparoscopic low anterior resection, left colectomy or right colectomy with an age of 16 years or older.

Exclusion Criteria:

* Duplicated data, subjects younger than 16, patients with previous abdominal surgery, and surgically complicated cases which were converted to open surgery were excluded.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study included all colorectal cancer patients over 2 years who were followed up or admitted to PSMMC under the service of colorectal surgery unit and who underwent laparoscopic low anterior resection, left colectomy or right colectomy with an age of 16 years or older.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Type of incision | Over 2 years
  The rate of incisional hernia development in relation to the incision site

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sultan Military Medical City, Riyadh, Saudi Arabia